CLINICAL TRIAL: NCT03469778
Title: Assessment of a Upper Limb Robotic Device in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 71611217.5.0000.0068
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2017-12

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; upper limb; motor activity; robotic
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic Therapy (Experimental): After consent, 10 participants will be included in a training program, as described below: 1º session will be robotic calibration and assessment; the following 18 sessions will be conducted the robotic therapy for upper limbs, three times a week. Each session will have a total duration of 55 minutes, including initial patient positioning and adjusting and after a sequence of game tasks.
  Interventions: Device: Robotic Therapy

INTERVENTIONS:
Device: Robotic Therapy — Robotic Therapy

SUMMARY:
The objectives of this phase II clinical study are: evaluate the efficacy, safety, patient adeherence and clinical applicability of a new robotic device for patients with stroke at a physical rehabilitation institution (Instituto de Medicina Física e Reabilitação do Hospital das Clínicas da Universidade de São Paulo - IMREA HCFMUSP - Rede de Reabilitação Lucy Montoro, unidade Vila Mariana). Methods: 10 patients with stroke diagnosis and Fugl-Meyer score ranging from 34 to 55 will be selected to be included in the study. After signing the informed consent form and being assessed by the baseline evaluations, they will undertake 18 sessions of robotic therapy, which in its turn will be prescribed three times a week. After this period, the patients will be evaluated for future comparison of both the pre-treatment and final assessments.

ELIGIBILITY:
Inlcusion Criteria:

1. Between 40 and 65 years.
2. Both genders.
3. Clinical and radiological diagnosis of ischemic stroke in the vascular territory of the middle cerebral artery or anterior cerebral artery.
4. Clinical assessment of disability with diagnosis of right or left hemiparesis.
5. Onset between 24 and 36 months.
6. Clinical stability verified in medical evaluation.
7. Spasticity less than or equal to 2 in Modified Ashworth Scale.
8. Moderate motor impairment in upper limb, according to Fugl-Meyer Assessment Upper Limb score (34 to 55 points).
9. To remain seated in a backrest chair during the intervention period (about 55 minutes).
10. Acceptance of informed consent form to participate in the study.

Exclusion Criteria:

1. Joint, muscle or tendinous lesions and/or pain that can occur during the intervention and make it difficult or impossible to perform robotic tasks.
2. Progressive worsening of spasticity.
3. Withdrawal of the informed consent form.
4. New episode of stroke.
5. Comorbidities that may occur during interventions such as hypertension, seizures, diabetes, among other uncontrolled clinical issues.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-05-02 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Assessment Upper Limb (FMA-UL) | Mean change from baseline at six weeks (19 sessions of robotic therapy).
  FMA-UL evaluates the recovery of the hemiplegic patient after stroke. It includes the measurement of reflex activity, movement with and without synergy, voluntary movements and coordination of shoulder, elbow, wrist, hand.

SECONDARY OUTCOMES:
Wolf Motor Function Test (WMFT) | Mean change from baseline at six weeks (19 sessions of robotic therapy).
  WMFT evaluates time performance and functional ability in 17 unimanual tasks.
Dynamometry - Grasp and Pinch | Mean change from baseline at six weeks (19 sessions of robotic therapy).
  Instrument to measure palmar and lateral grip (strength in kgf).
Patients safety | Adverse effects reported during 6 weeks treatment.
  Adverse effects questionnaire applied in each session.
Treatment adherence | Drop outs reported during 6 weeks treatment.
  Number of patients withdrawing from treatment without justification (drop outs).

OTHER OUTCOMES:
Clinical feasibility | Reported during 6 weeks treatment, in each session.
  Time necessary to adjust the device; patients satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Pesquisa Clínica - Instituto de Medicina Física e Reabilitação, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No